CLINICAL TRIAL: NCT00686361
Title: To Investigate Whether Choline Supplementation in Children With CF Will Correct Biochemical Markers of Choline Deficiency and Improve Plasma Indices of Methylation Capacity and Redox Status and Result in Decreased Pro-inflammatory Cytokines
Brief Title: Choline Nutrition in Children With Cystic Fibrosis (CF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Dr. Sheila M. Innis, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H06-70444
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; choline nutrition; choline and methyl metabolism; CF and oxidative stress
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Choline supplementation — Chart data, height, weight, pulmonary function, dietary intake and a venous blood and urine sample will be collected at enrollment then every 3 months for 9 months. Choline supplementation will be from enrollment for 6 months, with follow up at 3 months post supplementation. To avoid additional hospital visits and blood draws, and to co-ordinate with pulmonary function, hematology, clinical chemistry tests as part of clinical care, each subject will be seen at routine scheduled clinic appointments, which are every 3 months.

SUMMARY:
Cystic Fibrosis (CF) is a complex disease with a wide range of clinical problems. Despite enzyme replacement therapy, children with cystic fibrosis (CF) may still have problems absorbing some nutrients. Detailed studies of the nutrient status of children with CF and have found low amounts of choline, an essential dietary nutrient, and altered levels of some amino acids in almost all patients. Choline is an essential dietary nutrient that is important in many important body functions, which include proving a source of methyl groups, the structure of cell membranes and in acetylcholine. Most choline is present in our diets in a fat known as phosphatidylcholine. Research studies have shown that children with cystic fibrosis do not absorb fat, including phosphatidylcholine very well. In previous studies, we showed that choline provided as a dietary supplement for 2 weeks improved choline status in children with cystic fibrosis.

The purpose of this research is to find out if choline supplements over a longer duration of 6 months will improve and maintain normal choline status in children with CF.

DETAILED DESCRIPTION:
This is a prospective study involving 34 children attending an outpatient clinic for children with CF. After enrollment, subjects will be followed for 9 months with each child serving as their own control in a repeated measures design.

Chart data, height, weight, pulmonary function, dietary intake and a venous blood and urine sample will be collected at enrollment then every 3 months for 9 months. Choline supplementation will be from enrollment for 6 months, with follow up at 3 months post supplementation. To avoid additional hospital visits and blood draws, and to co-ordinate with pulmonary function, hematology, clinical chemistry tests as part of clinical care, each subject will be seen at routine scheduled clinic appointments, which are every 3 months.

The objectives are to

1. determine if supplementation with choline for 6 months corrects biochemical markers of choline deficiency and improves indices of reduced methylation capacity (including methionine, SAM, SAM/SAH) and redox status (GSH/GSSG) based on measures of blood and urine
2. determine whether or not choline supplementation decreases plasma pro-inflammatory mediators
3. determine if choline supplementation improves the low n-6 and n-3 fatty acids levels in children with CF,
4. explore if choline supplementation has the potential to have clinical relevance in reducing recurrent inflammation, and improve pulmonary function and/or reduce liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Children with Cystic Fibrosis of known genotype.

Exclusion Criteria:

* No hospitalizations within the previous month
* not receiving parenteral nutrition
* FEV1 > 50% at enrollment
* BMI and weight for age z-scores > 5th percentile
* non smokers
* no asthma
* not taking any lipid supplement or other agent designed to effect glutathione status.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Measured at: 0 (baseline), 3 and 6 mth (6 mth supplementation) and 9 mths (3 mth post supplementation) a) choline and methyl metabolites b) redox status (GSH/GSSG) | 9 months

SECONDARY OUTCOMES:
Measured at: 0, 3 and 6 mth and 9 mth a) inflammatory markers (IL-8, IL-6. IL-1ß, TNFα) b) essential n-6 and n-3 fatty acids c) pulmonary function (FVC, FEV1 (FEF 25-75) d) liver function (serum liver enzymes) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M. Innis, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Nutrition Research Program, BC Children's Hospital, Vancouver, British Columbia, Canada